CLINICAL TRIAL: NCT03274180
Title: A Prospective, Single-blind, Randomized Trial, of Non-inferiority of the Quality of Nurse Consultation Versus a Medical Consultation in Travel Medicine
Brief Title: Non-inferiority Trials of the Quality of Nurse Consultation Versus a Medical Consultation in Travel Medicine.
Acronym: aCTIVE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: K100104J
Record Dates: First submitted 2017-08-28; First posted 2017-09-06 (Actual); Last update posted 2017-09-28 (Actual); Status verified 2017-09

CONDITIONS: Travel and Motion
Keywords: Travel consultation

STUDY DESIGN:
Intervention Model Description: Experimental arm: Nurse consultation Non interventional arm: the medical consultation.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nursing consultation (Experimental): travel preventive consultation was performed by nurse
  Interventions: Other: Nursing consultation
- Medical consultation (No Intervention): travel preventive consultation was performed by a doctor

INTERVENTIONS:
Other: Nursing consultation — travel preventive consultation was performed by nurse
  Arms: Nursing consultation

SUMMARY:
A non inferiority mono-centre randomised single blind prospective study comparing a medical consultation versus nursing consultation, into two groups parallel without crossover.

DETAILED DESCRIPTION:
The permanent Survey of French data"monitoring of tourist demand" shows that 20% of the French population over 15 years performed each year at least one trip abroad. Travel most frequently are destined for European countries (6 times out of 10). The fact remains, however, that the french travelers (roughly 4.5 million) then fall between 120 countries of which a quarter part of the health high risk area.

Most of these risks can be minimized if appropriate precautions are observed before, during, and after the travel.

The development of tourism of people living in France is a real public health issue.

In these conditions, the need for travel medicine becomes more pressing. Medical discipline in full expansion, it is initially preventive before the trip. The other role of the travel medicine is the diagnosis and the treatment of the pathology after the end of the travel, which involves strictly medical skills.

This research investigation is so limited to travel preventive consultation before departure.

Regarding the prevention of the risks related to the trip, the World Health Organization (WHO) emits the 3 following recommendations:

"Travelers who intend to visit a developing country should consult a travel medicine center or a doctor, before their departure...". The main elements to look for by the healthcare professional who leads the consultation include:

* an assessment of any potential or underlying health problems
* a risk assessment linked to the trip according to destination, the route during the stay, the type of trip, the conditions and the duration of the stay
* the risk reduction strategy (Council in hygiene, nutrition) including the vaccinations and recommended therapeutics .

The consultation before the departure, interested on the promotion of health and the prevention of risks associated with travel. The aim is to propose suitable preventive measures. It cannot be a stereotyped speech depending on destinations, it is essential to adapt it to the person's situation.

Healthcare professionals must communicate effectively, so as to promote the understanding and retention of the information provided. The health promotion is one of the main skills invested by nurses.

The different investigation invites us to reflect on the new forms of health professionals cooperation. The investigator believe that the travel medicine offers opportunities in this way.

The hypothesis is : a nursing consultation in the travel medicine, subject to adequate training and a perfectly defined framework, can't meet the same criteria of quality of care than a medical consultation,

The expected results are an equivalence of results in terms of efficiency of support consultation.

ELIGIBILITY:
Inclusion Criteria:

* Traveler (male and female) over 18 years old (coming for travel consultation in a international center of vaccination)

Exclusion Criteria:

* Children and pregnant women,
* Travellers (man and woman) with co-morbidity factors as:

  * Hospitalization in the month previous consultation
  * Travelers with at least an one disease including an immune deficiency or dys-immunity, such as auto-immune disease,
  * Any recent discovery comorbidity (since less than 6 months)
  * Any traveler coming for consultation and bearer of signs of an acute health problem.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2017-09-25 (Actual); Primary Completion 2019-01-01 (Estimated); Study Completion 2019-08-01 (Estimated)

PRIMARY OUTCOMES:
Rate of memorization by travelers of the mains parameters related to the individual prevention of the traveler's Malaria, diarrhea and sexually transmitted infections. | At day 1
  Evaluated by a post-consultation memorization survey

SECONDARY OUTCOMES:
Quality score of the support consultation evaluating the memorization of Information by travelers. | At day 1
  Evaluated by memorisation survey
Level of satisfaction of travelers | At day 1
  The level of satisfaction will be assessed by a visual scale.
The relevance of the choice of vaccinations proposed in relation to recommendations | At day 1
  will be evaluated by a retrospective review
The relevance of the choice of prescribed anti-malarials in relation to recommendation | At day 1
  will be evaluated by a retrospective review

CONTACTS AND LOCATIONS:
Overall Officials: Delphine LECLERC, Nurse, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Service des Maladies Infectieuses et Tropicales, centre de conseils aux voyageurs, de vaccinations, Hôpital Avicenne, Bobigny, France

IPD SHARING:
Plan to Share IPD: No